CLINICAL TRIAL: NCT06749015
Title: A Multicenter, Retrospective, Observational Study on Treatment for Patients With BRAFV600E Mutant Metastatic Colorectal Cancer (mCRC)
Brief Title: A Study on Treatment for Patients With BRAFV600E Mutant Metastatic Colorectal Cancer (mCRC)
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiyu Chen, MD, PhD, Fudan University
Other Study IDs: BRAFm-mCRC
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer; BRAF V600 Mutation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No interventional: All BRAFV600E mutant patients having initiated treatment for mCRC between 01 October, 2020 and 01 October, 2025 (both days inclusive) with drugs registered for mCRC in respective study center
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
Previous studies have shown that BRAFV600E mutant mCRC patients have a shorter survival time than BRAF wild type mCRC patients. For Chinese patients, however, it remains unclear about the BRAF gene mutation rate, diagnosis, prognosis and survival data in people with BRAFV600E mutant mCRC .

This real-world, multicenter non-interventional study (NIS) will describe the mutation rate, treatment patterns, effectiveness and safety of current treatment regimens in BRAFV600E mutant mCRC patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed CRC that is metastatic and unresectable
* Presence of BRAFV600E mutation in tumor tissue, as confirmed by a local assay

Exclusion Criteria:

* patients with previous chronic inflammatory bowel disease, chronic diarrhea or recurrent bowel obstruction patients with symptomatic brain metastases active clinical severe infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis of histologically or cytologically confirmed mCRC with BRAFV600E mutation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 6 months
  the length of time between initiation of any line treatment for mCRC and the first documented disease progression

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  length of time between any treatment initiation (for mCRC) and death (due to any cause)
Overall Response rate (ORR) | 6 months
  number of complete response (CR) or partial response (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No